CLINICAL TRIAL: NCT03795805
Title: After Surgery Acute Renal Failure Incidence in Total Knee Arthroplasty With and Without Tourniquet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, JUAN LOPEZ VALENCIA, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R-2018-3401-053
Record Dates: First submitted 2018-12-26; First posted 2019-01-08 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Arthroplasty, Replacement, Knee; Acute Kidney Injury; Tourniquets; Knee Osteoarthritis
MeSH Terms: conditions — Acute Kidney Injury; Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee; Lidocaine

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TKA and Tourniquet (Other): Total knee arthroplasty and use of tourniquet limb cuff at 270 mmHg
  Interventions: Procedure: total knee arthroplasty; Procedure: Tourniquet limb cuff
- Intraarticular lidocain (Experimental): Total knee arthroplasty with Intaarticular lidocain
  Interventions: Procedure: total knee arthroplasty; Drug: Intaarticular lidocain

INTERVENTIONS:
Procedure: total knee arthroplasty — Total knee arhroplasty
  Other Names: TKA
Procedure: Tourniquet limb cuff — Tourniquet limb cuff and regular anesthesia
  Arms: TKA and Tourniquet
Drug: Intaarticular lidocain — 20 ml of 2% lidocain application intraarticular before surgery (intraarticular lidocain)
  Other Names: lidocaine
  Arms: Intraarticular lidocain

SUMMARY:
This study analize the incidence of acute renal failure after performing total knee arthroplasty with or without use of tourniquet limb cuff (half of patients for each group) in a randomized clinical trial

DETAILED DESCRIPTION:
This study analize the incidence of acute renal failure after performing total knee arthroplasty with or without (using local intraarticular anesthesia) use of tourniquet limb cuff (half of patients for each group) in a randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Patients knee arthrosis
* Required a surgical treatment with Total Knee Arthroplasty

Exclusion Criteria:

* Not accept to be in the study
* Not signed consent form
* Not having blood sample for creatinin meassure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Creatinin before surgery | Creatinin before surgery
  Blood Creatinin meassure in mg/dl before surgery
Creatinin after surgery 1 | Creatinin after surgery 1 at 24 hours
  Blood Creatinin meassure in mg/dl at 24 hours
Creatinin after surgery 2 | Creatinin after surgery 2 at 48 hours
  Blood Creatinin meassure in mg/dl at 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Avelino Colin Vázquez, MD, Principal Investigator — IMSS
Locations (1):
- UMAE Dr. Victorio de La Fuente Narvaez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
We will share only de demographic data and trial results